CLINICAL TRIAL: NCT04531332
Title: Efficacy and Safety of Continuous Infusion of Linezolid Compared With Intermittent Dosing in Critically Ill Pneumonic Patients
Brief Title: Continuous Infusion of Linezolid Versus Intermittent Dosing in the Treatment of Nosocomial Pneumonia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: October 6 University (Other)
Collaborators: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Ahmed Essam, Principle Investigator, October 6 University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-H-PhBSU-20004
Record Dates: First submitted 2020-07-30; First posted 2020-08-28 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Pneumonia
Keywords: linezolid continuous infusion; pneumonia; critically ill patients
MeSH Terms: conditions — Pneumonia | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuous infusion (Experimental): Patients will be received linezolid 600 mg intravenous Loading dose over 30 to 60 minutes followed by 1200 mg/ day by Continuous infusion (50 mg /hr)
  Interventions: Drug: Continuous infusion Linezolid
- Intermittent dosing (Active Comparator): Patients will be received Linezolid 600 mg intravenous twice daily over 30 to 60 minutes
  Interventions: Drug: intermittent dosing linezolid

INTERVENTIONS:
Drug: Continuous infusion Linezolid — Linezolid 600 mg intravenous Loading dose followed by 1200 mg/ day by Continuous infusion ( 50 mg /hr )
  Other Names: intervention
  Arms: Continuous infusion
Drug: intermittent dosing linezolid — Linezolid 600 mg intravenous twice daily
  Other Names: control
  Arms: Intermittent dosing

SUMMARY:
The investigator's goal in this study is to determine the clinical efficacy and safety of continuous infusion in comparison with standard intermittent infusion.

DETAILED DESCRIPTION:
Prospective randomized controlled clinical trial on critically ill Pneumonic patients, included two groups, over one year period. The first group will be administered intravenous (IV) linezolid 600mg twice daily. The second group will be prescribed linezolid (IV) 600 mg loading dose followed by 1200 mg by continuous infusion. Both groups will be co-administered intravenous (IV) Meropenem 1g every 8 hours empirically.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to ICUs diagnosed as HAP or VAP
* Chest X-ray/ computed tomography showing new or progressive infiltrate.
* New onset of purulent sputum or change in sputum character.
* Body temperature greater than 38 ℃ or less than 35.5℃.
* White blood cell counts greater than 10000 /mm3 or less than 4000 /mm3.
* Significant quantitative pathogen cultures from respiratory secretions.

Exclusion Criteria:

* Age <18 years, Pregnancy, Lactation
* Previous known allergic reaction to linezolid
* Creatinine Clearance (CrCl) <10 mL/min, calculated according to the Cockcroft-Gault formula
* Thrombocytopenia (platelet count less than 80,000/mm3)
* Severe hepatic failure (Child-Pugh C)
* Concomitant treatment with other drugs that can potentially interfere with Linezolid (i.e., macrolides, serotonin modulators, omeprazole)
* Acute DIC score > 4 points or hematological disorder
* Concurrent drug-associated Thrombocytopenia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult, Older Adult
Enrollment: 169 (Estimated)
Dates: Start 2019-11-15 (Actual); Primary Completion 2021-09-15 (Estimated); Study Completion 2021-09-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of cured patients in the linezolid continuous infusion group versus the proportion of cured patients in the intermittent group | through study completion, over one year
  The primary efficacy endpoint will be evaluated as clinical cure on day 7 of Linezolid initiation.
  Clinical cure defined by normalized body temperature, TLC less than 10,000/mL, absence of purulent secretions, and improvement of radiological findings (x-ray), in addition to Pao2/Fio2 greater than 250 in patients.
Percentage of occurrence of anemia and thrombocytopenia | through study completion, over one year
  The patients' hematological parameters (hemoglobin (Hb), hematocrit (Hct), and platelets (PLTs) counts) will be compared every 2 days during linezolid treatment between two groups.
  Anemia is defined as decrease in hemoglobin level <10 g/dl and Thrombocytopenia is defined as decrese in platelets count <100 × 103/mm3

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Essam, BSc, Principal Investigator — October 6 University
Locations (1):
- Beni-suef University, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No